CLINICAL TRIAL: NCT05718635
Title: Perforator Mapping and Optimizing Design of the Lateral Arm Flap: Clinical Trial
Brief Title: Perforator Mapping and Optimizing Design of the Lateral Arm Flap
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Osama Hassan Elbanna, Associate professor, Aswan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AswanU
Record Dates: First submitted 2022-10-12; First posted 2023-02-08 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Coverage of Soft Tissue Defects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients candidate for lateral arm flap (Experimental)
  Interventions: Diagnostic Test: coloured duplex; Procedure: supra facial dissection

INTERVENTIONS:
Diagnostic Test: coloured duplex — colored duplex to locate numbers sites and size of perforators.
Procedure: supra facial dissection — flap raising in supra facial plane

SUMMARY:
The goal of this clinical trial is to optimize the design of lateral arm flap. Colored duplex will be done for all Participants and compared to intra operative findings.

flap modification (Supra facial) dissection to lateral arm flap will be done and the results will compared to the ordinary method of dissection.

ELIGIBILITY:
Inclusion Criteria:

* adult patients

Exclusion Criteria:

* children injury to pedicle

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-03-26 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
numbers of perforators | two years
  numbers of perforators in the flap
site of perforators | two years
  distance from lateral humeral epicondyle in CM
Size of perforators | two years
  size in millimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided